CLINICAL TRIAL: NCT00324480
Title: A Phase I Study of Suberoylanilide Hydroxamic Acid (SAHA) in Combination With Flavopiridol in Advanced Solid Tumors
Brief Title: Vorinostat and Alvocidib in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00090; NCI-2009-00090 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MSKCC-05109; CDR0000472411; NCI-6858; 05-109 (Other: Memorial Sloan-Kettering Cancer Center); 6858 (Other: CTEP); P30CA008748 (NIH); U01CA069856 (NIH); NCT01645514 (obsolete NCT alias); NCT01664377 (obsolete NCT alias)
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2011-10

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — alvocidib; Vorinostat

ARMS (1):
- Treatment (chemotherapy, enzyme inhibitor) (Experimental): Before beginning course 1 of study therapy, patients receive oral SAHA on days 1-3 in order to ensure tolerability of the drug. Beginning 1 week later, patients receive oral SAHA once daily on days 1-3 and 8-10 and fixed-dose alvocidib IV over 1 hour on days 2 and 9. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvocidib; Drug: vorinostat; Other: pharmacological study

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat when given together with alvocidib in treating patients with advanced solid tumors. Drugs used in chemotherapy, such as vorinostat and alvocidib, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vorinostat together with alvocidib may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of vorinostat (SAHA) when given in combination with flavopiridol (alvocidib) in patients with advanced solid tumors.

II. Obtain preliminary data on the therapeutic activity of SAHA and flavopiridol in these patients.

III. Evaluate the role of p21, p53, and apoptotic markers relative to treatment response in patients treated with this regimen.

OUTLINE: This is a multicenter, open label, non-randomized, dose-escalation study of vorinostat (SAHA).

Before beginning course 1 of study therapy, patients receive oral SAHA on days 1-3 in order to ensure tolerability of the drug. Beginning 1 week later, patients receive oral SAHA once daily on days 1-3 and 8-10 and fixed-dose alvocidib intravenously (IV) over 1 hour on days 2 and 9. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 10 patients are treated at the MTD of SAHA in combination with fixed-dose alvocidib. Once the MTD of SAHA in combination with fixed-dose alvocidib is determined, patients receive oral SAHA at one dose level below the MTD once daily on days 1-3 and 8-10 and divided-dose alvocidib IV over 30 minutes followed by alvocidib IV over 4 hours on days 2 and 9. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. If this schedule is well-tolerated, the MTD of SAHA in combination with divided-dose flavopiridol is determined as above. An additional 10 patients are treated at the MTD of SAHA in combination with divided-dose alvocidib. Patients undergo blood draws on days 1 and 9 of course 1 for pharmacokinetic analysis.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor

  * Metastatic or unresectable disease
  * Standard curative or palliative measures do not exist or are no longer effective
* No hematologic malignancies
* No known brain metastases
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs
* No uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would preclude study compliance
* Recovered from prior therapy
* At least 2 weeks since prior histone acetylase inhibitors, including valproic acid
* At least 2 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* At least 2 weeks since prior investigational therapy
* At least 2 weeks since prior radiotherapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent commonly used vitamins, antioxidants, or herbal preparations and supplements

  * A single tablet multivitamin is allowed
* No other concurrent anticancer agents or therapies for this mailgnancy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-03; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of vorinostat when administered in combination with a fixed dose of weekly flavopiridol | Course 1
  Defined as the dose one level below the dose at which two or more of the patients in the initial cohort experience dose limiting toxicities (DLT) during the first treatment course. Graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 Term.

SECONDARY OUTCOMES:
Clinical pharmacokinetics of vorinostat (SAHA) | Week 1 of course 1
Therapeutic activity of SAHA and flavopiridol | Not Provided
Expression of p21, p53, and apoptotic markers relative to treatment response | Baseline to 2 weeks after completion of study treatment
  Evaluated using immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Schwartz, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States